CLINICAL TRIAL: NCT02620657
Title: A Retrospective Study on Real-world EGFR Mutation Testing Practice Status and Impact Factors in Patients With Advanced NSCLC in North China
Brief Title: Evaluate EGFR Mutation Status and Impact Factors in North China
Status: Completed | Type: Observational
Sponsor: ying cheng (Other)
Responsible Party: Sponsor-Investigator, ying cheng, Director of Jilin Cancer Hospital, Guangdong Association of Clinical Trials
Organization: Guangdong Association of Clinical Trials (Other)
Other Study IDs: 11224
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non interventional study: The patients with advanced NSCLC who have the medical records from Jan 1st 2014 to Dec 31st 2014 will be recruited .
  Interventions: Other: Non interventional study

INTERVENTIONS:
Other: Non interventional study — Non interventional study

SUMMARY:
Approximately 3000 advanced NSCLC patients, who fulfil the inclusion/exclusion criteria, will be recruited by 30 sites in North China.

DETAILED DESCRIPTION:
Approximately 3000 advanced NSCLC patients will be recruited , and the medical information of recruited patients must be recorded in the hospital electronic system from Jan 1st 2014 to Dec 31st 2014 .The study will focus on the EGFR testing rate in adenocarcinoma patients，so the collecting data for non-adenocarcinoma patients will be controlled in less than 10% for each site.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed NSCLC;
* Patients were diagnosed with advanced NSCLC from Jan 1st 2014 to Dec 31st 2014;
* Researchers should collect the records of consecutive NSCLC patients in each site.

Exclusion Criteria:

* Any patients without NSCLC diagnosis;
* Any patients which were diagnosed with advanced NSCLC before Jan 1st 2014 or after Dec 31st 2014.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 3000 advanced NSCLC patients
Sampling Method: Probability Sample
Enrollment: 2809 (Actual)
Dates: Start 2015-12; Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
To investigate the proportion of advanced NSCLC patients who performed EGFR mutation test | 2014.01.01-2014.12.31

CONTACTS AND LOCATIONS:
Overall Officials: CHENG NA Ying, Dr., Principal Investigator — Jilin Provincial Tumor Hospital

IPD SHARING:
Plan to Share IPD: No